CLINICAL TRIAL: NCT02178592
Title: ING117175: a Phase IIIb, Randomized, Open-label Study of the Safety and Efficacy of Dolutegravir or Efavirenz Each Administered With Two NRTIs in HIV-1-infected Antiretroviral Therapy-naïve Adults Starting Treatment for Rifampicin-sensitive Tuberculosis
Brief Title: Open-label Study of Dolutegravir (DTG) or Efavirenz (EFV) for Human Immunodeficiency Virus (HIV) - Tuberculosis (TB) Co-infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117175
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: integrase inhibitor; Mycobacterium tuberculosis; rifampicin-sensitive; dolutegravir; antiretroviral therapy-naïve; HIV-1 infection; efavirenz; co-infection
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections; Coinfection | interventions — dolutegravir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dolutegravir (Experimental): Twice-daily DTG 50 mg plus dual NRTI during RIF-containing TB treatment (isoniazid, RIF, pyrazinamide and ethambutol standard doses by the NTP under program conditions or acceptable alternative RIF-containing regimens) and for 2 weeks following discontinuation of TB treatment, then once-daily DTG 50 mg with the same NRTI through Week 52
  Interventions: Drug: DTG 50 mg
- Efavirenz (Active Comparator): Once-daily EFV 600 mg plus dual NRTI through Week 52 along with TB treatment including isoniazid, RIF, pyrazinamide and ethambutol standard doses by the NTP under program conditions.
  Interventions: Drug: EFV 600 mg

INTERVENTIONS:
Drug: DTG 50 mg — DTG is available as 50 mg film-coated tablet. DTG may be administered with or without food
  Arms: Dolutegravir
Drug: EFV 600 mg — EFV is supplied as film-coated capsule-shaped oral tablet containing 600 mg of EFV and must be administered without food
  Arms: Efavirenz

SUMMARY:
HIV/Tuberculosis (TB) co-infection have profound effects on the host's immune system. TB is the most common cause of death in patients with HIV worldwide. Rifamycins (such as rifampicin [RIF]) are an important component of TB therapy because of their unique activity. The problem is that most protease inhibitors (PI) and non-nucleoside reverse transcriptase inhibitors (NNRTI) used to treat HIV have significant drug-drug interactions with RIF that can lead to reduced concentrations of these agents with risk of treatment failure or resistance. The non-nucleoside reverse transcriptase inhibitor (NNRTI) efavirenz (EFV) does not present the same significant drug interactions with RIF. EFV-based HIV treatment was tested in patients concomitantly treated with RIF-containing TB therapy, demonstrating that their co-administration can be used safely and effectively. However, the side effect profile of EFV overlaps with the RIF-containing TB regimens and makes the management of treatment toxicities very complex. Integrase inhibitors (INI), such as dolutegravir (DTG), may offer an important alternative to EFV-based therapy in TB coinfected patients. A Phase I drug-drug interaction study was conducted in healthy, HIV-seronegative subjects, and showed that DTG at 50 mg twice daily given together with RIF was well-tolerated and resulted in DTG concentrations similar to those of DTG 50 mg given once daily alone, which is the recommended dose for INI-naive patients. Therefore, ART regimens using DTG 50 mg twice daily may represent a new treatment option for TB-infected patients who require concurrent treatment for HIV infection. This is a Phase III b, randomized, open-label study describing the efficacy and safety of DTG and EFV-containing ART regimens in HIV/TB co-infected patients. This study is designed to assess the antiviral activity of DTG or efavirenz (EFV) ART-containing regimens through 48 weeks. A total of approximately 115 +/-5% subjects will be randomly assigned in a 3:2 ratio to DTG (approximately 69 subjects) and EFV (approximately 46 subjects), respectively. This study will include a Screening Period, a Randomized Phase (Day 1 to 48 weeks plus a 4-week extension), and a DTG Open-label extension (OLE). During the DTG OLE, subjects will be supplied with DTG until it is locally approved and commercially available, the subject no longer derives clinical benefit, or the subject meets a protocol-defined reason for discontinuation, which ever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Subject or the subject's legal representative is willing and able to understand and provide signed and dated written informed consent prior to Screening
* Adult subject (at least 18 years of age) with plasma HIV-1 RNA>=1000 copies/ milliliter (mL) at Screening
* CD4+ cell count is >= 50 cells/ cubic millimetre (mm^3) at Screening
* HIV-1-infected, ART-naïve; (<=10 days of prior therapy with any antiretroviral drug following a diagnosis of HIV-1 infection)
* A female subject may be eligible to enter and participate in the study if she: is of non-childbearing potential defined as either postmenopausal (12 months of spontaneous amenorrhea and >=45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy, or bilateral oophorectomy or, is of childbearing potential, with a negative pregnancy test at both Screening and Day 1, and agrees to use one of the following methods of contraception to avoid pregnancy
* Complete abstinence from intercourse from 2 weeks prior to administration of IP, throughout the study, and for at least 2 weeks after discontinuation of all study medications
* Double-barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide)
* Approved hormonal contraception plus a barrier method while receiving Rifampicin (RIF)-containing TB treatment for subjects randomly assigned to the DTG arm or approved hormonal contraception plus a barrier method for subjects randomly assigned to the EFV arm (regardless of RIF-containing TB treatment)
* Any intrauterine device with published data showing that the expected failure rate is <1% per year
* Male partner sterilization prior to the female subject's entry into the study and this male is the sole partner for that subject
* Any other method with published data showing that the expected failure rate is <1% per year
* Any contraception method must be used consistently, in accordance with the approved product label and for at least 2 weeks after discontinuation of study drug. A childbearing potential female subject who starts the study using complete abstinence as her contraceptive method and decides to become sexually active must use the double barrier method either as a bridge to an approved hormonal contraception (if possible) or as a method of choice to be maintained from that moment onwards
* All subjects participating in the study should be counseled on safer sexual practices including the use of effective barrier methods
* New diagnosis of pulmonary, pleural, or Lymph node (LN) TB based on identification of Mycobacterium tuberculosis using culture methods or validated nucleic acid amplification test on sputum or on samples collected by needle aspirate of pleural fluid or an affected LN
* RIF sensitivity of Mycobacterium tuberculosis either by culture or validated nucleic acid amplification test
* RIF-containing first-line TB treatment or an alternate RIF-containing TB treatment started up to a maximum of 8 weeks before randomization and no later than the screening date
* Karnofsky score >=70% before randomization

Exclusion Criteria:

* Any previous TB treatment (not including treatment for latent disease)
* Evidence of RIF resistance of Mycobacterium tuberculosis either by culture or validated nucleic acid amplification test
* Expected requirement for TB treatment >9 months
* Concomitant disorders or conditions for which isoniazid, RIF, pyrazinamide, or ethambutol are contraindicated
* Central nervous system, miliary, or pericardial TB
* Women who are pregnant or breastfeeding
* Any evidence of an active Acquired immunodeficiency syndrome (AIDS)-defining disease (Centers for Disease Control and Prevention, Category C). Exceptions include TB, cutaneous Kaposi's sarcoma not requiring systemic therapy, and historic CD4+ cell counts of <200 cells/mm^3
* Subjects with moderate to severe hepatic impairment (Class B or C) as determined by Child-Pugh classification unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Subjects positive for hepatitis B surface antigen (HBsAg) at screening
* Anticipated need for hepatitis C virus (HCV) therapy during the Randomized Phase of the study
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the investigator and the study medical monitor for inclusion of the subject
* Subjects who, in the investigator's judgment, pose a significant suicidality risk. Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any of the following agents within 28 days of Screening: radiation therapy, cytotoxic chemotherapeutic agents, any immunomodulators that alter immune response
* Treatment with any agent, other than licensed ART as allowed above with documented activity against HIV-1 in vitro/vivo within 28 days of first dose of IP
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of IP
* Any evidence of primary viral resistance to Nucleoside reverse transcriptase inhibitor (NRTIs), Non-nucleoside reverse transcriptase inhibitor (NNRTIs), or Protease inhibitor (PIs) based on the presence of any major resistance-associated mutation (according to the International AIDS Society Update of the Drug Resistant Mutations in HIV-1 ) in the Screening result or, if known, any historical resistance test result. Note: Retests of Screening genotypes are not allowed
* Any verified Grade 4 laboratory abnormality
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the subject's participation in the study of an investigational compound
* Alanine aminotransferase >=2 × upper limit of normal
* Hemoglobin <=7.4 grams per deciliter;
* Platelet count <50000/mm^3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-01-23 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (23):
- Argentina (2):
  - GSK Investigational Site, Ciudad de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
- Brazil (4):
  - GSK Investigational Site, Manaus, Amazonas
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, DF
- Peru (3):
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Iquitos, Loreto
  - GSK Investigational Site, Lima
- Russia (2):
  - GSK Investigational Site, Oryol
  - GSK Investigational Site, Saint Petersburg
- South Africa (7):
  - GSK Investigational Site, Soweto, Gauteng
  - GSK Investigational Site, Durban, KwaZulu-Natal
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Klerksdorp
  - GSK Investigational Site, Observatory, Cape Town
  - GSK Investigational Site, Westdene
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen

REFERENCES:
- [Background] Dooley KE, Kaplan R, Mwelase N, Grinsztejn B, Ticona E, Lacerda M, Sued O, Belonosova E, Ait-Khaled M, Angelis K, Brown D, Singh R, Talarico CL, Tenorio AR, Keegan MR, Aboud M; International Study of Patients with HIV on Rifampicin ING study group. Dolutegravir-based Antiretroviral Therapy for Patients Coinfected With Tuberculosis and Human Immunodeficiency Virus: A Multicenter, Noncomparative, Open-label, Randomized Trial. Clin Infect Dis. 2020 Feb 3;70(4):549-556. doi: 10.1093/cid/ciz256. PMID 30918967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 7 countries across 25 centers; Argentina (2), Brazil (4), Mexico (3), Peru (4), Russia (2), South Africa (8) and Thailand (2). Participants were randomized to receive either Dolutegravir (DTG) or Efavirenz (EFV) containing regimens.
Pre-assignment Details: A total of 263 participants were screened of which 150 were screen failures. A total of 113 participants were enrolled in this study.
Groups:
- DTG 50 mg: Participants in this arm received DTG 50 milligrams (mg) tablet with or without food twice-daily with 2 Nucleoside Reverse Transcriptase Inhibitors (NRTIs), Tuberculosis (TB) treatment including isoniazid, rifampicin (RIF), pyrazinamide, and ethambutol provided at standard doses by the National TB Control Program (NTP) under program conditions until 2 weeks after TB therapy was completed and then received DTG 50 mg once daily (with the same NRTI backbone) through the end of the Randomized Phase up to Week 52. Participants continued receiving DTG 50 mg once daily during the open-label extension phase (OLE) until DTG became locally approved and commercially available to all participating countries (occurred up to Week 252).
- EFV 600 mg: Participants in this arm received EFV 600 mg tablet administered without food plus 2 NRTIs (TB treatment including isoniazid, RIF, pyrazinamide, and ethambutol provided at standard doses by the NTP under program conditions) through the end of the Randomized Phase up to Week 52. All participants receiving EFV then left the study and transitioned to locally-available EFV, except for participants randomized to EFV in South Africa who completed 2 years within the OLE phase and transitioned to locally available EFV regimens or withdrew from study prior to transitioning to locally-available EFV.
Period: Randomized Phase (Up to Week 52)
Arm/Group | DTG 50 mg | EFV 600 mg
Started | 69 | 44
Completed | 50 | 35
Not Completed | 19 | 9
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 11 | 3
Not completed — Physician Decision | 1 | 0
Period: OLE Phase (Week 52 to Week 252)
Arm/Group | DTG 50 mg | EFV 600 mg
Started | 47 (As OLE phase was optional, 3 participants from DTG arm did not enter OLE from Randomized Phase.) | 19 (As OLE phase was optional, 16 participants from EFV arm did not enter OLE from Randomized Phase.)
Completed | 35 | 16
Not Completed | 12 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Reached Protocol defined stopping criteria | 2 | 0
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG 50 mg | EFV 600 mg | Total
Number analyzed (Participants) | 69 | 44 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (10.25) | 33.1 (7.56) | 34.0 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 16 | 46
  Male | 39 | 28 | 67
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 47 | 28 | 75
  American Indian or Alaska Native | 11 | 4 | 15
  Asian - South East Asian Heritage | 0 | 2 | 2
  White - Arabic/North African Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 9 | 9 | 18
  Mixed Race | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) < 50 Copies/Milliliter at Week 48 in DTG Arm Using the Modified United States (US) Food and Drug Administration (FDA) Snapshot Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The percentage of participants with plasma HIV-1 RNA <50 copies/milliliter was assessed at Week 48 using the snapshot algorithm in the DTG arm. Response was assessed using a modified FDA Snapshot algorithm in which participants were not penalized for any single protocol allowed background therapy substitution even if occurs after the first trial visit. In this approach participants with HIV-1 RNA >=50 copies/milliliter are considered as non-responders. Participants without HIV-1 RNA data at Week 48 (due to missing data or discontinuation of investigational product [IP] prior to visit window) are also considered as non-responders, as well as participants with anti-retroviral (ART) substitutions were not permitted. Study drug (i.e. DTG or EFV) was not allowed to be substituted.
Time Frame: Week 48
Population: Intent-to-treat exposed (ITT-E) Population comprised of all randomly assigned participants who received at least one dose of IP.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG 50 mg
Number analyzed (Participants) | 69
Percentage of participants | 75 [65 to 86]

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/Milliliter at Week 48 in EFV Arm Using the Modified Snapshot Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The percentage of participants with plasma HIV-1 RNA <50 copies/milliliter were assessed at Week 48 using the snapshot algorithm in the EFV arm. Response was assessed using a modified FDA Snapshot algorithm in which participants were not penalized for any single protocol allowed background therapy substitution even if occurs after the first trial visit. In this approach participants with HIV-1 RNA >=50 copies/milliliter are considered as non-responders. Participants without HIV-1 RNA data at Week 48 (due to missing data or discontinuation of IP prior to visit window) are also considered as non-responders, as well as participants with ART substitutions were not permitted. Study drug (i.e. DTG or EFV) was not allowed to be substituted.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | EFV 600 mg
Number analyzed (Participants) | 44
Percentage of participants | 82 [70 to 93]

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 Copies/Milliliter at Week 24 in Both EFV and DTG Arms Using the Modified Snapshot Algorithm
Description: Plasma samples were collected for quantitative analysis of HIV-1 RNA. The percentage of participants with plasma HIV-1 RNA <50 copies/milliliter were assessed at Week 24 using the snapshot algorithm in the DTG and EFV arm. Response was assessed according to the Modified Snapshot algorithm. In this approach participants with HIV-1 RNA >=50 copies/milliliter were considered non-responders. Participants without HIV-1 RNA data at Week 24 (due to missing data or discontinuation of IP prior to visit window) were also considered as non-responders, as well as participants with ART substitutions were not permitted. Substitution of a background NRTI agent was permissible one time if it was due to reasons of drug toxicity.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Percentage of participants | 81 [72 to 90] | 89 [79 to 98]

4. Secondary Outcome: Percentage of Participants Without Confirmed Virologic Withdrawal and Without Discontinuation Due to Treatment-related Reasons at Week 24 and Week 48
Description: Percentage of participants not meeting confirmed virologic withdrawal criteria nor discontinued due to treatment related reasons at the time of analysis at Week 24 (through Day 210) and Week 48 (through Day 350) has been presented by treatment group. The time to meeting confirmed virologic withdrawal criteria or discontinuation due to treatment related reasons (i.e., discontinuation due to drug-related adverse event [AE], or due to protocol defined safety stopping criteria, or due to lack of efficacy) were calculated. Participants who met confirmed virologic withdrawal criteria or discontinuation due to treatment related reasons were considered as Failure. Participants who had not met confirmed virologic withdrawal criteria (per protocol) and were ongoing in the study, or who had discontinued for reasons other than those related to treatment, were censored. This would be the Treatment-Related Discontinuation = Failure (TRDF) data.
Time Frame: Week 24 and Week 48
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Percentage of participants
  Week 24 | 98.4 [89.1 to 99.8] | 95.2 [82.1 to 98.8]
  Week 48 | 96.6 [87.0 to 99.1] | 92.7 [79.1 to 97.6]

5. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Counts at Week 24 and Week 48
Description: Blood samples were collected for assessment of lymphocyte subsets (CD4+ lymphocyte count) by flow cytometry at Baseline and Weeks 24, 48. Baseline was defined as the last pre-treatment value observed (typically from Day 1 visit). Change from Baseline was calculated subtracting the value at the specified time point from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: ITT-E Population. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Cells per millimeter^3
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Cells per millimeter^3
  Week 24, n=61,41: number analyzed (Participants) | 61 | 41
  Week 24, n=61,41 | 153.2 (125.09) | 127.1 (158.14)
  Week 48, n=49, 33: number analyzed (Participants) | 49 | 33
  Week 48, n=49, 33 | 199.0 (146.22) | 194.5 (137.81)

6. Secondary Outcome: Number of Participants With Serious Adverse Event (SAE) and Common (>=5%) Non-serious AE (Non-SAE) - Randomized Phase
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward medical occurrence that, at any dose that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, all events of possible drug-induced liver injury with hyperbilirubinemia or any other situation according to medical or scientific judgment. Data for number of participants with SAE and common (>=5%) non-SAE over 52 weeks has been summarized.
Time Frame: Up to Week 52
Population: Safety Population comprised of all participants who received at least one dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Participants
  Common Non-SAE | 38 | 33
  SAE | 5 | 5

7. Secondary Outcome: Number of Participants With SAE and Common (>=5%) Non-SAE - OLE Phase
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward medical occurrence that, at any dose that results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, all events of possible drug-induced liver injury with hyperbilirubinemia or any other situation according to medical or scientific judgment. Data for number of participants with SAE and common (>=5%) non-SAE from Week 52 to Week 252 has been summarized.
Time Frame: Week 52 to Week 252
Population: Safety OLE Population comprised of all participants in Safety Population who entered the OLE phase.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 47 | 19
Participants
  Common Non-SAE | 36 | 16
  SAE | 5 | 2

8. Secondary Outcome: Number of Participants With Maximum Post-Baseline-emergent Chemistry Toxicities - Randomized Phase
Description: Blood samples for assessment of clinical chemistry parameters were collected at indicated time points. Clinical chemistry assessments included alanine aminotransferase (ALT), albumin, alkaline phosphatase, aspartate aminotransferase (AST), bilirubin, carbon dioxide, cholesterol, creatine kinase, creatinine, glucose, low density lipoprotein (LDL) cholesterol calculation, lipase, phosphate, potassium, and sodium. Data for number of participants who experienced maximum post-Baseline emergent chemistry toxicities were summarized. Maximum post-Baseline emergent chemistry toxicities were graded using Division of Acquired Immune Deficiency Syndrome (DAIDS) toxicity grading for HIV-infected participants as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life-threating). Higher grade indicates more severity.
Time Frame: Up to Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Participants
  ALT, Grade 1 | 10 | 9
  ALT, Grade 2 | 1 | 1
  ALT, Grade 3 | 1 | 1
  ALT, Grade 4 | 0 | 0
  Albumin, Grade 1 | 2 | 2
  Albumin, Grade 2 | 8 | 1
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  Alkaline phosphatase, Grade 1 | 7 | 11
  Alkaline phosphatase, Grade 2 | 0 | 1
  Alkaline phosphatase, Grade 3 | 0 | 0
  Alkaline phosphatase, Grade 4 | 0 | 0
  AST, Grade 1 | 11 | 8
  AST, Grade 2 | 4 | 3
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 1 | 1
  Bilirubin, Grade 1 | 3 | 3
  Bilirubin, Grade 2 | 1 | 0
  Bilirubin, Grade 3 | 0 | 0
  Bilirubin, Grade 4 | 0 | 0
  Carbon dioxide, Grade 1 | 14 | 8
  Carbon dioxide, Grade 2 | 4 | 4
  Carbon dioxide, Grade 3 | 1 | 0
  Carbon dioxide, Grade 4 | 0 | 0
  Cholesterol, Grade 1 | 5 | 6
  Cholesterol, Grade 2 | 1 | 2
  Cholesterol, Grade 3 | 0 | 0
  Cholesterol, Grade 4 | 0 | 0
  Creatine kinase, Grade 1 | 3 | 4
  Creatine kinase, Grade 2 | 0 | 0
  Creatine kinase, Grade 3 | 0 | 0
  Creatine kinase, Grade 4 | 1 | 1
  Creatinine, Grade 1 | 2 | 0
  Creatinine, Grade 2 | 0 | 0
  Creatinine, Grade 3 | 0 | 1
  Creatinine, Grade 4 | 0 | 0
  Glucose, Grade 1 | 11 | 10
  Glucose, Grade 2 | 3 | 5
  Glucose, Grade 3 | 0 | 0
  Glucose, Grade 4 | 0 | 0
  LDL cholesterol calculation, Grade 1 | 0 | 3
  LDL cholesterol calculation, Grade 2 | 1 | 0
  LDL cholesterol calculation, Grade 3 | 0 | 0
  LDL cholesterol calculation, Grade 4 | 0 | 0
  Lipase, Grade 1 | 2 | 2
  Lipase, Grade 2 | 0 | 2
  Lipase, Grade 3 | 0 | 0
  Lipase, Grade 4 | 0 | 1
  Phosphate, Grade 1 | 5 | 3
  Phosphate, Grade 2 | 3 | 5
  Phosphate, Grade 3 | 1 | 0
  Phosphate, Grade 4 | 0 | 0
  Potassium, Grade 1 | 5 | 3
  Potassium, Grade 2 | 0 | 2
  Potassium, Grade 3 | 0 | 0
  Potassium, Grade 4 | 1 | 1
  Sodium, Grade 1 | 17 | 9
  Sodium, Grade 2 | 2 | 3
  Sodium, Grade 3 | 1 | 0
  Sodium, Grade 4 | 0 | 0

9. Secondary Outcome: Number of Participants With Maximum Post-Baseline-emergent Chemistry Toxicities- Randomized Phase + OLE Phase
Description: Blood samples for assessment of clinical chemistry parameters were collected at indicated time points. Clinical chemistry assessments included ALT, albumin, alkaline phosphatase, AST, bilirubin, carbon dioxide, cholesterol, creatine kinase, creatinine, glucose, LDL cholesterol calculation, lipase, phosphate, potassium, and sodium. Data for number of participants with maximum post-Baseline emergent chemistry toxicities were summarized. Maximum post-Baseline emergent chemistry toxicities were graded using DAIDS toxicity grading for HIV-infected participants as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life-threating) . Higher grade indicates more severity.
Time Frame: Up to Week 252
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Participants
  ALT, Grade 1 | 12 | 10
  ALT, Grade 2 | 3 | 2
  ALT, Grade 3 | 1 | 1
  ALT, Grade 4 | 0 | 0
  Albumin, Grade 1 | 2 | 2
  Albumin, Grade 2 | 8 | 1
  Albumin, Grade 3 | 0 | 0
  Albumin, Grade 4 | 0 | 0
  Alkaline phosphatase, Grade 1 | 8 | 12
  Alkaline phosphatase, Grade 2 | 0 | 1
  Alkaline phosphatase, Grade 3 | 0 | 0
  Alkaline phosphatase, Grade 4 | 0 | 0
  AST, Grade 1 | 14 | 8
  AST, Grade 2 | 6 | 3
  AST, Grade 3 | 1 | 1
  AST, Grade 4 | 1 | 1
  Bilirubin, Grade 1 | 7 | 3
  Bilirubin, Grade 2 | 1 | 0
  Bilirubin, Grade 3 | 0 | 0
  Bilirubin, Grade 4 | 0 | 0
  Carbon dioxide, Grade 1 | 16 | 10
  Carbon dioxide, Grade 2 | 5 | 4
  Carbon dioxide, Grade 3 | 1 | 0
  Carbon dioxide, Grade 4 | 0 | 0
  Cholesterol, Grade 1 | 5 | 6
  Cholesterol, Grade 2 | 1 | 2
  Cholesterol, Grade 3 | 0 | 0
  Cholesterol, Grade 4 | 0 | 0
  Creatine kinase, Grade 1 | 7 | 4
  Creatine kinase, Grade 2 | 1 | 1
  Creatine kinase, Grade 3 | 0 | 0
  Creatine kinase, Grade 4 | 2 | 1
  Creatinine, Grade 1 | 2 | 0
  Creatinine, Grade 2 | 1 | 0
  Creatinine, Grade 3 | 0 | 1
  Creatinine, Grade 4 | 0 | 0
  Glucose, Grade 1 | 12 | 12
  Glucose, Grade 2 | 7 | 5
  Glucose, Grade 3 | 0 | 0
  Glucose, Grade 4 | 0 | 0
  LDL cholesterol calculation, Grade 1 | 0 | 3
  LDL cholesterol calculation, Grade 2 | 1 | 0
  LDL cholesterol calculation, Grade 3 | 0 | 0
  LDL cholesterol calculation, Grade 4 | 0 | 0
  Lipase, Grade 1 | 3 | 2
  Lipase, Grade 2 | 0 | 3
  Lipase, Grade 3 | 0 | 0
  Lipase, Grade 4 | 0 | 1
  Phosphate, Grade 1 | 5 | 5
  Phosphate, Grade 2 | 10 | 7
  Phosphate, Grade 3 | 1 | 1
  Phosphate, Grade 4 | 0 | 0
  Potassium, Grade 1 | 8 | 3
  Potassium, Grade 2 | 0 | 2
  Potassium, Grade 3 | 0 | 0
  Potassium, Grade 4 | 1 | 1
  Sodium, Grade 1 | 22 | 9
  Sodium, Grade 2 | 3 | 3
  Sodium, Grade 3 | 1 | 0
  Sodium, Grade 4 | 0 | 0

10. Secondary Outcome: Number of Participants With Maximum Post-Baseline-emergent Hematology Toxicities- Randomized Phase
Description: Blood samples for assessment of hematology parameters were collected at indicated time points. Hematology assessments included hemoglobin, leukocytes, neutrophils and platelets. Data for number of participants who experienced maximum post-Baseline emergent hematology toxicities were summarized. Maximum post-Baseline emergent hematology toxicities were graded using DAIDS toxicity grading for HIV-infected participants as Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe) and Grade 4 (potentially life-threating). Higher grade indicates more severity.
Time Frame: Up to Week 52
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Participants
  Hemoglobin, Grade 1 | 2 | 1
  Hemoglobin, Grade 2 | 0 | 0
  Hemoglobin, Grade 3 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grade 1 | 4 | 1
  Leukocytes, Grade 2 | 0 | 0
  Leukocytes, Grade 3 | 0 | 1
  Leukocytes, Grade 4 | 0 | 1
  Neutrophils, Grade 1 | 6 | 3
  Neutrophils, Grade 2 | 2 | 1
  Neutrophils, Grade 3 | 1 | 0
  Neutrophils, Grade 4 | 1 | 2
  Platelets, Grade 1 | 2 | 1
  Platelets, Grade 2 | 0 | 0
  Platelets, Grade 3 | 1 | 0
  Platelets, Grade 4 | 0 | 0

11. Secondary Outcome: Number of Participants With Maximum Post-Baseline-emergent Hematology Toxicities - Randomized Phase + OLE Phase
Description: as for outcome 10
Time Frame: Up to Week 252
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Participants
  Hemoglobin, Grade 1 | 2 | 1
  Hemoglobin, Grade 2 | 1 | 0
  Hemoglobin, Grade 3 | 0 | 0
  Hemoglobin, Grade 4 | 0 | 0
  Leukocytes, Grade 1 | 5 | 3
  Leukocytes, Grade 2 | 1 | 1
  Leukocytes, Grade 3 | 0 | 1
  Leukocytes, Grade 4 | 0 | 1
  Neutrophils, Grade 1 | 4 | 2
  Neutrophils, Grade 2 | 5 | 3
  Neutrophils, Grade 3 | 2 | 0
  Neutrophils, Grade 4 | 2 | 3
  Platelets, Grade 1 | 0 | 2
  Platelets, Grade 2 | 1 | 0
  Platelets, Grade 3 | 2 | 0
  Platelets, Grade 4 | 0 | 0

12. Secondary Outcome: Percent Change From Baseline in the Fasting Lipid Profile at Week 24 and Week 48
Description: Samples for lipid measurements were obtained in a fasted state at Baseline, Week 24 and Week 48. The parameters assessed during the lipid profile were total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, triglycerides. Baseline was defined as the last pre-treatment value observed (typically from Day 1 visit). Percent change from Baseline for a parameter was calculated as the observed value minus the Baseline value divided by Baseline value multiplied by 100. Data for fasting lipid parameters has been summarized.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented as n=X in the category titles). Data for this outcome measure has been presented until Week 48 only (Randomized Phase) as per protocol. It was not planned for OLE Phase, hence data was not collected for OLE Phase.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Percent change
  Cholesterol, Week 24, n=58, 40: number analyzed (Participants) | 58 | 40
  Cholesterol, Week 24, n=58, 40 | 6.314 (20.7036) | 16.443 (22.0445)
  Cholesterol, Week 48, n=47, 34: number analyzed (Participants) | 47 | 34
  Cholesterol, Week 48, n=47, 34 | -0.375 (21.4890) | 17.371 (20.6312)
  HDL Cholesterol, Week 24, n=58, 40: number analyzed (Participants) | 58 | 40
  HDL Cholesterol, Week 24, n=58, 40 | 39.002 (53.5060) | 39.174 (49.1087)
  HDL Cholesterol, Week 48, n=47, 34: number analyzed (Participants) | 47 | 34
  HDL Cholesterol, Week 48, n=47, 34 | 24.987 (48.2471) | 45.423 (52.9949)
  LDL Cholesterol, Week 24, n=58, 40: number analyzed (Participants) | 58 | 40
  LDL Cholesterol, Week 24, n=58, 40 | 4.315 (31.7095) | 13.487 (36.2511)
  LDL Cholesterol, Week 48, n=47, 34: number analyzed (Participants) | 47 | 34
  LDL Cholesterol, Week 48, n=47, 34 | -2.957 (31.9910) | 9.132 (41.1942)
  Triglycerides, Week 24, n=58, 40: number analyzed (Participants) | 58 | 40
  Triglycerides, Week 24, n=58, 40 | -22.744 (33.4148) | 16.934 (118.7319)
  Triglycerides, Week 48, n=47, 34: number analyzed (Participants) | 47 | 34
  Triglycerides, Week 48, n=47, 34 | -18.402 (39.0227) | 13.175 (57.0389)

13. Secondary Outcome: Change From Baseline in the Fasting Lipid Profile for Total Cholesterol/HDL Ratio at Week 24 and Week 48
Description: Samples for lipid measurements were obtained in a fasted state at Baseline, Week 24 and Week 48. The parameter assessed during the lipid profile was total cholesterol/HDL ratio. Baseline was defined as the last pre-treatment value observed (typically from Day 1 visit). Change from baseline for a parameter was calculated as the observed value minus the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 48
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Ratio of total cholesterol to HDL
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Ratio of total cholesterol to HDL
  Total cholesterol/HDL ratio, Week 24, n=58, 40: number analyzed (Participants) | 58 | 40
  Total cholesterol/HDL ratio, Week 24, n=58, 40 | -16.292 (22.7982) | 36.562 (315.0478)
  Total cholesterol/HDL ratio, Week 48, n=47, 34: number analyzed (Participants) | 47 | 34
  Total cholesterol/HDL ratio, Week 48, n=47, 34 | -11.949 (27.5044) | -11.051 (28.3183)

14. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Study Treatment Due to AEs - Randomized Phase
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Data for percentage of participants who permanently discontinued study treatment due to any AE over 52 weeks has been summarized.
Time Frame: Up to Week 52
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 69 | 44
Percentage of participants | 0 | 5

15. Secondary Outcome: Percentage of Participants Who Permanently Discontinued Study Treatment Due to AEs - OLE Phase
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Data for percentage of participants who permanently discontinued study treatment due to any AE from Week 52 to Week 252 has been summarized.
Time Frame: Week 52 to Week 252
Population: Safety OLE Population
Measure: Number; unit: Percentage of participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 47 | 19
Percentage of participants | 4 | 0

16. Secondary Outcome: Number of Participants With Tuberculosis (TB) Associated (Assoc.) Immune Reconstitution Inflammatory Syndrome (IRIS)
Description: Participants were monitored for signs and symptoms of TB-assoc. IRIS. Participants with IRIS symptoms in any AE or HIV assoc. conditions were classified by Endpoint Adjudication Committee in following four categories: met criteria for TB-assoc. IRIS, possibly met criteria for TB-assoc. IRIS, suspected TB-assoc. IRIS but not possible to adjudicate and No TB associated IRIS. They were further graded from Grades 1 to 4 using DAIDS. Higher grade indicates more severity. The preliminary requirements to meet TB-assoc. IRIS criteria were diagnosis of TB and initial response to TB treatment (stabilized or improved condition of participant in presence of TB treatment before starting ART). The clinical criteria was onset of IRIS signs and symptoms related to TB should occur within first 3 months of starting, restarting or changing ART regimen for treatment failure. Number of participants who sent to the adjudication committee and analyzed were presented.
Time Frame: Up to Week 12
Population: Safety Population. Only those participants with data available at the specified time points were analyzed. Data for this outcome measure has been presented until Week 12 only (Randomized phase) as per protocol. It was not planned for OLE Phase, hence data was not collected for OLE Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 9 | 12
Participants
  Met criteria for TB-assoc. IRIS, Grade 1 | 1 | 0
  Met criteria for TB-assoc. IRIS, Grade 2 | 2 | 3
  Met criteria for TB-assoc. IRIS, Grade 3 | 1 | 0
  Met criteria for TB-assoc. IRIS, Grade 4 | 0 | 1
  Possibly met criteria for TB-assoc. IRIS, Grade 1 | 0 | 0
  Possibly met criteria for TB-assoc. IRIS, Grade 2 | 0 | 0
  Possibly met criteria for TB-assoc. IRIS, Grade 3 | 0 | 0
  Possibly met criteria for TB-assoc. IRIS, Grade 4 | 0 | 0
  Suspected TB-assoc. IRIS unable to adjudicate, Grade 1 | 0 | 0
  Suspected TB-assoc. IRIS unable to adjudicate, Grade 2 | 0 | 0
  Suspected TB-assoc. IRIS unable to adjudicate, Grade 3 | 0 | 0
  Suspected TB-assoc. IRIS unable to adjudicate, Grade 4 | 0 | 0
  No TB associated IRIS | 5 | 8

17. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance
Description: Whole venous blood samples were obtained from each participant until Week 52 for potential viral genotypic and phenotypic analyses. Genotypic and phenotypic testing was conducted for participants meeting confirmed virologic withdrawal criteria, i.e., confirmed HIV-1 RNA >=400 copies/milliliter from Week 24 onwards. Genotypic and phenotypic analyses was carried out by Monogram Biosciences using, but not limited to, their Standard Phenosense and GenoSure testing methods for protease (PRO), reverse transcriptase (RT), and integrase assays. Data for number of participants with treatment-emergent genotypic resistance mutations have been presented for the RT region on codons G190G, K101K, K103K, K65K, V106V and Y181Y.
Time Frame: Up to Week 52
Population: Viral Genotypic Population comprised of all participants in the ITT-E Population with available on-treatment genotypic data at the time confirmed virologic withdrawal was met.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 2 | 1
Participants
  G190G (wild type) | 2 | 0
  G190G/A | 0 | 1
  K101K (wild type) | 2 | 0
  K101K/E | 0 | 1
  K103K (wild type) | 2 | 0
  K103K/N | 0 | 1
  K65K (wild type) | 2 | 0
  K65R | 0 | 1
  V106V (wild type) | 2 | 0
  V106M | 0 | 1
  Y181Y (wild type) | 2 | 0
  Y181Y/C | 0 | 1

18. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance
Description: Phenotypic susceptibility to all licensed antiretroviral drugs, including DTG and EFV were determined using PhenoSense HIV assays from Monogram Inc. Clinical cutoffs or biological cutoffs by PhenoSense were used to define the phenotypic susceptibility of background treatment and were interpreted as fold change > clinical lower cut-off or biologic cut-off as resistance, fold change <=clinical lower cut-off or biologic cut-off as sensitive, and fold change > clinical higher cut-off as resistance, fold change <=clinical higher cut-off and > clinical lower cut-off as partially sensitive, and fold change <=clinical lower cut-off as sensitive. Data has been presented for participants with treatment-emergent phenotypic resistance.
Time Frame: Up to Week 52
Population: Viral Phenotypic Population comprised of all participants in the ITT-E Population with available on-treatment phenotypic resistance data at the time confirmed virologic withdrawal criteria was met. Only participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | DTG 50 mg | EFV 600 mg
Number analyzed (Participants) | 2 | 1
Participants
  Dolutegravir, Sensitive, n=1,1: number analyzed (Participants) | 1 | 1
  Dolutegravir, Sensitive, n=1,1 | 1 | 1
  Dolutegravir, Partially sensitive, n=1,1: number analyzed (Participants) | 1 | 1
  Dolutegravir, Partially sensitive, n=1,1 | 0 | 0
  Dolutegravir, Resistance, n=1,1: number analyzed (Participants) | 1 | 1
  Dolutegravir, Resistance, n=1,1 | 0 | 0
  Elvitegravir, Sensitive, n=1,1: number analyzed (Participants) | 1 | 1
  Elvitegravir, Sensitive, n=1,1 | 1 | 1
  Elvitegravir, Resistance, n=1,1: number analyzed (Participants) | 1 | 1
  Elvitegravir, Resistance, n=1,1 | 0 | 0
  Raltegravir, Sensitive, n=1,1: number analyzed (Participants) | 1 | 1
  Raltegravir, Sensitive, n=1,1 | 1 | 1
  Raltegravir, Resistance, n=1,1: number analyzed (Participants) | 1 | 1
  Raltegravir, Resistance, n=1,1 | 0 | 0
  Delavirdine, Sensitive, n=2,1 | 2 | 1
  Delavirdine, Resistance, n=2,1 | 0 | 0
  Efavirenz, Sensitive, n=2,1 | 2 | 0
  Efavirenz, Resistance, n=2,1 | 0 | 1
  Etravirine, Sensitive, n=2,1 | 2 | 1
  Etravirine, Partially sensitive, n=2,1 | 0 | 0
  Etravirine, Resistance, n=2,1 | 0 | 0
  Nevirapine, Sensitive, n=2,1 | 2 | 0
  Nevirapine, Resistance, n=2,1 | 0 | 1
  Rilpivirine, Sensitive, n=2,1 | 2 | 1
  Rilpivirine, Resistance, n=2,1 | 0 | 0
  Abacavir, Sensitive, n=2,1 | 2 | 1
  Abacavir, Partially sensitive, n=2,1 | 0 | 0
  Abacavir, Resistance, n=2,1 | 0 | 0
  Didanosine, Sensitive, n=2,1 | 2 | 0
  Didanosine, Partially sensitive, n=2,1 | 0 | 0
  Didanosine, Resistance, n=2,1 | 0 | 1
  Emtricitabine, Sensitive, n=2,1 | 2 | 0
  Emtricitabine, Resistance, n=2,1 | 0 | 1
  Lamivudine, Sensitive, n=2,1 | 2 | 0
  Lamivudine, Resistance, n=2,1 | 0 | 1
  Stavudine, Sensitive, n=2,1 | 2 | 1
  Stavudine, Resistance, n=2,1 | 0 | 0
  Tenofovir, Sensitive, n=2,1 | 2 | 0
  Tenofovir, Partially sensitive, n=2,1 | 0 | 1
  Tenofovir, Resistance, n=2,1 | 0 | 0
  Zidovudine, Sensitive, n=2,1 | 2 | 1
  Zidovudine, Resistance, n=2,1 | 0 | 0
  Atazanavir, Sensitive, n=2,1 | 2 | 1
  Atazanavir, Resistance, n=2,1 | 0 | 0
  Darunavir, Sensitive, n=2,1 | 2 | 1
  Darunavir, Partially sensitive, n=2,1 | 0 | 0
  Darunavir, Resistance, n=2,1 | 0 | 0
  Fosamprenavir, Sensitive, n=2,1 | 2 | 1
  Fosamprenavir, Partially sensitive, n=2,1 | 0 | 0
  Fosamprenavir, Resistance, n=2,1 | 0 | 0
  Indinavir,Sensitive, n=2,1 | 2 | 1
  Indinavir, Resistance, n=2,1 | 0 | 0
  Lopinavir, Sensitive, n=2,1 | 2 | 1
  Lopinavir, Partially sensitive, n=2,1 | 0 | 0
  Lopinavir, Resistance, n=2,1 | 0 | 0
  Nelfinavir, Sensitive, n=2,1 | 2 | 1
  Nelfinavir, Resistance, n=2,1 | 0 | 0
  Ritonavir, Sensitive, n=2,1 | 2 | 1
  Ritonavir, Partially sensitive, n=2,1 | 0 | 0
  Ritonavir, Resistance, n=2,1 | 0 | 0
  Saquinavir, Sensitive, n=2,1 | 2 | 1
  Saquinavir, Partially sensitive, n=2,1 | 0 | 0
  Saquinavir, Resistance, n=2,1 | 0 | 0
  Tipranavir, Sensitive, n=2,1 | 2 | 1
  Tipranavir, Partially sensitive, n=2,1 | 0 | 0
  Tipranavir, Resistance, n=2,1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-SAEs were collected up to Week 52 for Randomized Phase and from Week 52 to Week 252 for OLE Phase.
Description: Safety Population was used to assess SAEs and non-SAEs for Randomized Phase which comprised of all participants who received at least one dose of IP. Safety OLE Population was used to assess SAEs and non-SAEs for OLE Phase which comprised of all participants in Safety Population who entered the OLE phase. AEs were presented treatment-wise and phase-wise.
Groups:
- DTG 50 mg- Randomized Phase: In randomized phase, participants received DTG 50 mg tablet with or without food twice-daily with 2 NRTIs, TB treatment including isoniazid, RIF, pyrazinamide, and ethambutol provided at standard doses by the NTP under program conditions until 2 weeks after TB therapy was completed and then received DTG 50 mg once daily (with the same NRTI backbone) through 52 weeks.
- EFV 600 mg- Randomized Phase: In randomized phase, participants received EFV 600 mg tablet administered without food plus 2 NRTIs, TB treatment including isoniazid, RIF, pyrazinamide, and ethambutol provided at standard doses by the NTP under program conditions through 52 weeks.
- DTG 50 mg- OLE Phase: In OLE Phase, participants received DTG 50 mg tablet until DTG became locally approved and commercially available.
- EFV 600 mg- OLE Phase: In OLE Phase, participants received EFV 600 mg tablet.
Arm/Group | DTG 50 mg- Randomized Phase | EFV 600 mg- Randomized Phase | DTG 50 mg- OLE Phase | EFV 600 mg- OLE Phase
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/44 | 1/47 | 0/19
Serious Adverse Events (participants affected / at risk) | 5/69 | 5/44 | 5/47 | 2/19
Other Adverse Events (participants affected / at risk) | 38/69 | 33/44 | 36/47 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50 mg- Randomized Phase (N=69) | EFV 600 mg- Randomized Phase (N=44) | DTG 50 mg- OLE Phase (N=47) | EFV 600 mg- OLE Phase (N=19)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Tuberculosis gastrointestinal (Infections and infestations) | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Hypocalcaemic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DTG 50 mg- Randomized Phase (N=69) | EFV 600 mg- Randomized Phase (N=44) | DTG 50 mg- OLE Phase (N=47) | EFV 600 mg- OLE Phase (N=19)
Upper respiratory tract infection (Infections and infestations) | 5 | 8 | 12 | 5
Lower respiratory tract infection (Infections and infestations) | 9 | 3 | 4 | 3
Pharyngitis (Infections and infestations) | 5 | 3 | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 5 | 3 | 2
Herpes zoster (Infections and infestations) | 3 | 3 | 0 | 0
Body tinea (Infections and infestations) | 4 | 0 | 1 | 1
Headache (Nervous system disorders) | 9 | 6 | 5 | 4
Dizziness (Nervous system disorders) | 3 | 6 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 10 | 4 | 3
Vomiting (Gastrointestinal disorders) | 5 | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 4 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 3 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 4 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 3 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 3 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Tinea faciei (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis gastrointestinal (Infections and infestations) | 0 | 0 | 0 | 1
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 0
Blood pressure increased (Investigations) | 4 | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02178592/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT02178592/SAP_003.pdf